CLINICAL TRIAL: NCT06403891
Title: The Effect of a Comprehensive Rehabilitation Program Using Robotic Walking and Functional Electrical Stimulation Technologies on Balance and Walking in Children With Cerebral Palsy
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-22-1398
Record Dates: First submitted 2024-04-24; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: The control group was planned to consist of patients who received a 6-week conventional rehabilitation program that was prepared to meet the requirements of their clinical conditions, including neurophysiological exercises, balance-coordination and posture exercises.
- Case: The case group was planned to consist of patients who received a comprehensive rehabilitation program using high-tech devices including functional electrical stimulation (FES) and robotic rehabilitation applications in addition to the conventional rehabilitation program that was prepared to meet the requirements of their clinical conditions, including neurophysiological exercises, balance-coordination and posture exercises.

SUMMARY:
The aim of this study was to investigate the effect of a comprehensive rehabilitation program using robotic walking and functional electrical stimulation technologies on balance and gait in children with cerebral palsy. This study was planned as a prospective observational study. A total of 30 patients in two groups were planned to be included in the study. Patients in both groups were planned to receive a 6-week conventional rehabilitation program that was prepared to meet the requirements of their clinical conditions, including neurophysiological exercises, balance-coordination and posture exercises. The case group was planned to consist of patients who received a comprehensive rehabilitation program using high-tech devices including functional electrical stimulation (FES) and robotic rehabilitation applications in addition to the conventional rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 2-18
* Being diagnosed with cerebral palsy
* Walking independently with or without an assistive walking device
* Having a GMFCS score between 1-3
* Lack of seizure history
* Showing consent to participate in the study (signing the informed consent by the legal guardian of the patient)

Exclusion Criteria:

* Presence of contracture in lower extremities
* Being administered botulinum toxin within the last one month before treatment or during the 6-week treatment period
* Being unable to cooperate with clinical assessments

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients between the ages of 2-18, diagnosed with cerebral palsy, receiving inpatient treatment in Ankara Bilkent City Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Cadence | The first assessment was planned before the rehabilitation program, and the second assessment was planned at the end of the 6-week rehabilitation program
  The number of steps taken per minute
Step length | The first assessment was planned before the rehabilitation program, and the second assessment was planned at the end of the 6-week rehabilitation program
  The distance between the initial contact of one foot and the initial contact of the contralateral foot
Stride length | The first assessment was planned before the rehabilitation program, and the second assessment was planned at the end of the 6-week rehabilitation program
  The distance between the consecutive initial contacts of the same foot
Track width | The first assessment was planned before the rehabilitation program, and the second assessment was planned at the end of the 6-week rehabilitation program
  The mediolateral distance between right and left heels during gait
Range of motion of joints during the gait cycle | The first assessment was planned before the rehabilitation program, and the second assessment was planned at the end of the 6-week rehabilitation program
  Range of motion of the knee, hip and ankle joint during the gait cycle
Range of motion of the pelvis in the frontal plane during the gait cycle | The first assessment was planned before the rehabilitation program, and the second assessment was planned at the end of the 6-week rehabilitation program
  Range of motion of the pelvis in the frontal plane during the gait cycle
Plantar surface pressure distribution | The first assessment was planned before the rehabilitation program, and the second assessment was planned at the end of the 6-week rehabilitation program
  Plantar surface pressure distribution measured by pedobarograph

SECONDARY OUTCOMES:
Spasticity | The first assessment was planned before the rehabilitation program, and the second assessment was planned at the end of the 6-week rehabilitation program
  Spasticity will be assessed with the Modified Ashworth Scale
Balance | The first assessment was planned before the rehabilitation program, and the second assessment was planned at the end of the 6-week rehabilitation program
  Balance will be assessed with the Pediatric Berg Balance Scale
Gait speed | The first assessment was planned before the rehabilitation program, and the second assessment was planned at the end of the 6-week rehabilitation program
  Gait speed will be assessed with the 10-meter walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)